CLINICAL TRIAL: NCT05070962
Title: Complex Post-traumatic Stress Disorder: What Symptomatological Specificities
Acronym: StuCoTra
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Raincy Montfermeil Hospital Group (Network)
Responsible Party: Sponsor
Other Study IDs: GHT_ CHIRB -RIPH2_003
Record Dates: First submitted 2021-09-14; First posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Psychiatric Health
Keywords: Disorder,; complex post-traumatic stress disorder; personality disorders
MeSH Terms: conditions — Disease; Personality Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical population: having experienced repeated and prolonged traumatic exposure
  Interventions: Other: clinical population
- General population: Student volunteers from the University of Lille
  Interventions: Other: clinical population

INTERVENTIONS:
Other: clinical population — or the general population, students of the University of Lille will be offered the opportunity to participate in a study through posters in the corridors of the faculties and announcements in the lecture halls.
  Other Names: general poupulation

SUMMARY:
A better understanding of the Complex Post-Traumatic Stress Disorder would allow a management as close as possible to the specificities of this one, but also a better training of professionals and adapted therapeutic indications.

DETAILED DESCRIPTION:
Post-Traumatic Stress Disorder manifests itself in a multitude of symptoms and self-regulation difficulties in various domains (somatization and biological balance, attention and consciousness, regulation of affects and impulses, interpersonal relationships and relational capacities, perception of the aggressor and of the aggression, self-perception and identity, sense and belief system) as well as profound changes in personality and various comorbidities .In addition, dissociation, the origin and the resulting disorders also have some similarities to Complex Post-Traumatic Stress Disorder. Indeed, dissociation is thought to have a traumatic origin and the symptomatology (eg hyperesthesia, dissociative amnesia, anesthesia) is included in Complex Post-Traumatic Stress Disorder. We can then ask ourselves the following questions: is Complex Post-Traumatic Stress Disorder a dissociative disorder in its own right causing difficulties with self-regulation? What is the share of dissociation in Complex Post-Traumatic Stress Disorder?

ELIGIBILITY:
Inclusion Criteria:

For clinical population;

* Age between 18 and 65 years old;
* Having experienced repeated and prolonged traumatic exposure;
* Able to understand and answer self-questionnaires;
* Having expressed their free and informed consent
* Affiliated with a social security scheme

For general population:

* Student volunteers from the University of Lille;
* Aged between 18 and 65 years old;
* Able to understand and answer self-questionnaires;
* Having expressed their free and informed consent.

Exclusion Criteria:

For clinical population;

* People with difficulties in answering the self-questionnaires (e.g. incomprehension of items, emotional difficulties);
* Persons under tutorship or curatorship;
* Persons deprived of their liberty.

For general population:

* People with difficulties in answering the self-questionnaires (e.g. incomprehension of items, emotional difficulties);
* Persons under tutorship or curatorship;
* Persons deprived of their liberty;
* Persons having a link of subordination with the investigative team.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The clinical population is made up of individuals who are victims of repeated trauma and are cared for in specialized centers; The general reference population is made up of volunteer students from the University of Lille.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-02-17 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
the symptomatological characteristics of Complex Post-Traumatic Stress Disorder | during the study
  to evaluate the symptomatic characteristics of TSPTc evoked by the authors (cognitions, emotional regulation, comorbidities, etc.) in order to better identify the symptomatic specificities of the disorder and improve its management.

SECONDARY OUTCOMES:
Validation of the French version of two self-assessment scales; | during the study
  Validate the French-language version of two TSPTc self-assessment scales (SIDES-SR and ITQ) on a French population;
differences in self-assessment of the participant's overall functioning and personality | during the study
  differences in participant's general functioning and personality self-assessment between tCPD and personality disorders - specifically Borderline Personality Disorder (BPD).

CONTACTS AND LOCATIONS:
Overall Officials: Marion SIMION, Principal Investigator — USAP CHI Robert Ballanger
Locations (1):
- USAP CHI Robert Ballanger Boulevard Robert Ballanger, Aulnay-sous-Bois, France

IPD SHARING:
Plan to Share IPD: No